CLINICAL TRIAL: NCT01831947
Title: Efficacy of Ranibizumab Treatment Every 2 Month Compared to Treatment on Demand on Patients With Choroidal Neo-vascularization (CNV) as a Consequence of Age-related Macular Degeneration (AMD)
Brief Title: Efficacy Study of Ranibizumab on Patients With Age-related Macular Degeneration.
Acronym: RABIMO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other)
Collaborators: Novartis Pharmaceuticals (Industry); University Medical Center Goettingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002ADE09T
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Macular Degeneration
Keywords: age-related macular degeneration; Ranibizumab
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab fixed dose (Experimental): Injection of 0.5 mg Ranibizumab every 2 months for one year, following a monthly injection during the first 3 months.
  Interventions: Biological: Ranibizumab
- Ranibizumab on demand (Experimental): Injection of 0.5 mg Ranibizumab on demand for one year, following a monthly injection during the first 3 months.
  Interventions: Biological: Ranibizumab

INTERVENTIONS:
Biological: Ranibizumab
  Other Names: Lucentis (Novartis Pharma)

SUMMARY:
This clinical trial investigates the impact of intravitreal injection of Ranibizumab antibody on the acuteness of vision. Patients included are suffering from choroidal neo-vascularization (CNV) as a consequence of age-related macular degeneration (AMD).

Initially, all patients get injections of 0.5 mg Ranibizumab in monthly intervals for 3 months. Subsequently, one group gets Ranibizumab in intervals of 2 months, whereas a second group is treated on demand.

The primary end point of the study is the change of best-corrected visual acuity after 12 month.

Secondary end points include the impact of Ranibizumab on morphological changes of the retina, the number of patients with gain or loss of 15 or more letters visual acuity after 12 months, changes in quality of life and the number of injections required during the first 12 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with choroidal neo-vascularization (CNV) as a consequence of age-related macular degeneration (AMD)
* age 50 and older, male and female
* membrane <= 12 papillary diameter
* visual acuity between 20/320 and 20/40 (ETDRS)
* written informed consent

Exclusion Criteria:

* known hypersensitivity to the medicinal product under investigation, ingredients or medicinal products with a similar chemical structure
* participation in another clinical trial within the last 4 weeks
* unability to understand trial information
* pregnant or lactating women
* women with an amenorrhea < 12 months
* suspected unability to cooperate
* detachment of pigment epithelium without membrane detection >= 50%,retinal angiomatotic proliferation (RAP), presumed ocular histoplasmosis syndrome (POHS), chorioretinal anastomosis (CRA), myopic CNV, CNV following trauma, uveitis, RCS or reasons except AMD
* rupture of pigment epithelium
* sub-retinal bleeding >= 50% of membrane or >= 1 PD
* sub-retinal fibrosis or chorio-atrophy
* pre-treatment with Verteporfin (photodynamic therapy), radiotherapy, trans-pupillary thermotherapy of the eye under investigation as a consequence of maculadegeneration treatment with Verteporfin of the eye not under investigation within 7 days prior inclusion
* former participation in clinical trials with anti-angiogenic substances: Pegaptanib, Ranibizumab, Bevacizumab, Anecortave Acetat, Proteinkinase C Inhibitors
* former injection of anti-angiogenic substances in the eye under investigation
* former focal sub-foveal lasercoagulation of the eye under investigation
* juxta- or extra-foveal lasercoagulation of the eye under investigation within 1 month prior inclusion
* former vitrectomy
* former surgery as a consequence of maculadegeneration
* glaucoma patients which have been treated with prostaglandin containing eye drops
* other ocular diseases which may lead to surgery within the clinical study or may lead to a loss of vision of two lines
* acute intraocular inflammation of the eye under investigation
* vitreous hemorrhage of the eye under investigation
* macula-foramen of the eye under investigation
* diabetic retinopathy
* former retina detachment of the eye under investigation
* uveitis
* acute conjunctivitis, keratitis, scleritis, or endophthalmitis
* aphakia or pseudo-aphakia with damaged back-capsule(exception: YAG-capsulotomy)
* myopia larger than -8 diopter
* former intra-ocular surgery of the eye under investigation within 2 months prior inclusion
* de-compensated glaucoma with >= 30 mm Hg despite therapy
* former filtrating glaucoma surgery of the eye under investigation
* former corneal grafting of the eye under investigation
* former stroke or heart attack
* on-going therapy because of systemic infection
* known allergic reaction to fluorescein
* bad quality of fundus documentation because of bad range of vision

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
best-corrected visual acuity | 12 months after start of treatment
  Change of best-corrected visual acuity before and 12 months after start of treatment with respect to number of letters read on ETDRS-sheets (Early Treatment Diabetes Retinopathy Study Sheets).

SECONDARY OUTCOMES:
Fluoresceinangiography | 12 months after start of treatment
  To study morphological and anatomical changes of the retina. Affected area is determined in mm²
Photography | 12 months after treatment start
  To study morphological and anatomical changes of the retina. Affected area is assessed by computer-assisted measurement in mm².
optical coherence tomography (OCT) | 12 months after treatment start
  To study morphological and anatomical changes of the retina. Thickness of the retina is determined in µm².
number of injections | 12 months after treatment start
quality of life | 12 months after treatment start
  change in quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Ophthalmology, University Medical Center Goettingen, Göttingen, Germany